CLINICAL TRIAL: NCT06146712
Title: A Single-Group Study to Examine the Efficacy of a Melatonin Lotion With Magnesium to Improve Sleep Quality and Quantity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asutra (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20360
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm: 'Dream the night away' nighttime lotion (Experimental): The product should be applied once daily at night (30 minutes before bedtime). Participants should apply two teaspoons (one teaspoon of lotion covers approximately the size of the fingertip from tip to first knuckle) of lotion (3 mg of melatonin) and use it wherever they would usually use body lotion (paying particular attention to areas of tension in shoulders, neck, and temples, or on their legs and feet if they experience restless legs or muscle tightness).
  Participants should do this for 20 nights.
  Interventions: Other: Asutra's 'Dream the night away' nighttime lotion

INTERVENTIONS:
Other: Asutra's 'Dream the night away' nighttime lotion — Product contains Water (Aqua), Magnesium Chloride, Dimethyl Sulfone (MSM), Prunus Amygdalus Dulcis (Sweet Almond) Oil, Butyrospermum Parkii (Shea Butter), Sodium Lactate, Cetearyl Alcohol, Glyceryl Stearate Citrate, Glycerin, Undecane, Cetyl Palmitate, Polyglyceryl-3 Diisostearate, Pentylene Glycol, Glyceryl Stearate, Magnesium Sulfate, Melatonin, Tridecane, Potassium Chloride, Sodium Chloride, Calcium Chloride, Tocopheryl Acetate, Xanthan Gum, Hydroxyacetophenone, Sodium Hydroxide, Cymbopogon Flexuosus (East-Indian Lemongrass) Oil, Citral, Geraniol, Linalool

SUMMARY:
This study will evaluate the efficacy of Asutra's 'Dream the night away' nighttime lotion with melatonin and magnesium on sleep health in terms of quantity, quality, ease of falling asleep or falling back asleep after waking in the night, and grogginess upon waking. The study will be conducted as a virtual single-group trial in which all 35 participants will use the test product. This study will last 3 weeks, and participants will use the product daily (each night 30 minutes before bedtime for 20 nights). Participants will use a sleep tracker to monitor their sleep for a week at Baseline (before commencing the trial) and nightly throughout the trial. Participants will complete study-specific questionnaires at Baseline, and after first use, 3 days, 1 week, 2 weeks, and 3 weeks, in which they will also record the results from their sleep tracker.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-59.
* Must agree to not use any other sleep aids including prescriptions, supplements, or melatonin products during the study or 28 days prior to Baseline.
* Has favorable sleep conditions (a dark, quiet room to sleep in and is not woken up regularly throughout the night due to personal circumstances e.g. by a baby).
* Willing to maintain their standard sleep pattern and activity level for the duration of the study.
* Be generally healthy and not living with any uncontrolled chronic disease. Willing and able to supply and use their own sleep tracking device.

Exclusion Criteria:

* Diagnosed with any chronic sleep condition including insomnia, narcolepsy, or sleep apnea.
* Has extremely sensitive/irritable skin or diagnosed skin conditions.
* Has poor sleep hygiene as a result of specific personal circumstances e.g. new mothers.
* Women who are pregnant, breastfeeding, or attempting to become pregnant.
* Anyone unwilling or unable to follow the study protocol.
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Is currently undergoing, or planning to to undergo any sleep-related procedures in the next three weeks.
* A history of severe allergic reactions including but not limited to any of the product's ingredients.
* Heavy drinkers or drug users. A heavy drinker is considered to be a woman who drinks 8 or more alcoholic drinks per week or a man who drinks 15 or more alcoholic drinks per week.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Changes in scores on the validated Sleep Quality Scale (SQS). [Timeline: Baseline to Week 3] | 3 weeks
  Consisting of 28 items, the SQS evaluates six domains of sleep quality: daytime symptoms, restoration after sleep, problems initiating. Using a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "some- times," 2 = "often," and 3 = "almost always").
Changes in time asleep recorded by a wearable sleep tracker. [Timeline: Baseline to Week 3] | 3 weeks
  The total time asleep every night will be recorded using a wearable sleep tracker, the Fitbit Inspire 3.
Changes in "sleep score" given by wearable sleep tracker. [Timeline: Baseline to Week 3] | 3 weeks
  The Fitbit Inspire 3 gives a nightly "sleep score". This is based on heart rate, the time spent awake or restless, and the sleep stages. The score is out of 100, with 100 being the best possible score.

SECONDARY OUTCOMES:
Participants' perceptions of the product's efficacy. [Timeline: Baseline to Week 3] | 3 weeks
  Participants' perception of the product's efficacy in improving sleep quality will be assessed via study-specific questionnaire. Participants will respond to Likert-scale questions (0-4 point scale) with 0=the least favourable score and 4=the most favourable score.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided